CLINICAL TRIAL: NCT06842173
Title: Randomized, Double-Blind, Placebo-Controlled Phase I/II Clinical Trial To Evaluate The Safety And Immunogenicity Of The Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) From Instituto Butantan, In Adults And The Older Adults
Brief Title: Safety and Immunogenicity of the Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented and Adjuvanted) in Adults and Older Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Fundação Butantan (Unknown); Butantan Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLP-02-IB
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Avian Influenza A Virus
Keywords: Influenza A Virus Subtype H5N8; Avian Influenza; Safety; Immunogenicity
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Intervention Model Description: Double-blind clinical trial. Randomization, preparation and masking of the Product Under Investigation by an unblinded professional at the research site.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monovalent Influenza Vaccine A (H5N8) 7.5 mcg (Experimental): Intervention: Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) from Instituto Butantan, containing 7.5 mcg/dose of hemagglutinin (HA) and adjuvant IB160 (0.5 mL/dose of final combined product).
  Interventions: Biological: Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) 7.5 mcg
- Monovalent influenza vaccine A (H5N8) 15 mcg (Experimental): Intervention: Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) from Instituto Butantan, containing 15 mcg/dose of hemagglutinin (HA) and adjuvant IB160 (0.5 mL/dose of final combined product).
  Interventions: Biological: Monovalent influenza vaccine type A (H5N8) 15 mcg
- Placebo (Placebo Comparator): Phosphate buffered saline (PBS) (0.5 mL/dose).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) 7.5 mcg — Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) 7.5 mcg + IB160 adjuvant (0.5mL total)
  Other Names: Avian Flu vaccine
  Arms: Monovalent Influenza Vaccine A (H5N8) 7.5 mcg
Biological: Monovalent influenza vaccine type A (H5N8) 15 mcg — Monovalent influenza vaccine type A (H5N8) 15 mcg + IB160 adjuvant (0.5mL total)
  Other Names: Avian Flu vaccine
  Arms: Monovalent influenza vaccine A (H5N8) 15 mcg
Other: Placebo — Phosphate buffered saline (PBS) (0.5 mL/dose).
  Other Names: Control arm
  Arms: Placebo

SUMMARY:
This study aims to demonstrate the safety and immunogenicity of two formulations of the monovalent influenza vaccine candidate A (H5N8) (inactivated, fragmented, and adjuvanted with IB160) from the Instituto Butantan in adults and older adults, to be developed for situations of pandemic, epidemic or outbreak of avian type A/H5 in humans, in the context of pandemic preparedness.

DETAILED DESCRIPTION:
This is a clinical trial (randomized, double-blind, placebo-controlled Phase I/II) to evaluate the safety and immunogenicity of two formulations of the monovalent influenza vaccine candidate A (H5N8) (inactivated, fragmented, and adjuvanted with IB160) from the Instituto Butantan in adults and older adults. Safety will be assessed by the frequency (n, %) of participants with solicited (local and systemic) and unsolicited adverse events reported within 7 days post each vaccination; as well as the frequency of adverse reactions post causality evaluation. Immunogenicity will be assessed by seroprotection and seroconversion rates in the 21 days after the second dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females aged ≥ 18 years at the time of the first study vaccination.
2. Be in good health and clinically stable (defined as having no pre-existing health condition or having a pre-existing health condition that has not required a change in treatment or hospitalization for worsening of disease in the 3 months prior to the date of the first study vaccination).
3. Agree to participate in the study and provide written informed consent prior to the initiation of any study procedures.
4. Be able and willing to comply with all study procedures, including completing Participant Diaries, collecting blood samples, and being available for scheduled study visits and contacts.
5. For females of childbearing potential, have a negative pregnancy test prior to the first study vaccination.
6. For women of childbearing potential, be willing to use effective contraceptive measures during the screening visit until at least 30 days after the second study vaccination.

Exclusion Criteria:

1. Having received any vaccine (including seasonal influenza) 28 days prior to the date of the first study vaccination or having any vaccination in the period from the first vaccination to the immune response assessment visit after the last vaccination.
2. Known hypersensitivity or allergy to eggs, chicken proteins, squalene-based adjuvants, or any other component of the investigational product.
3. History of serious adverse reaction or anaphylaxis to any previous influenza vaccine (licensed or not).
4. Having received any influenza A/H5 vaccine or history of exposure to avian influenza A/H5.
5. Presence of a bleeding disorder or any condition that contraindicates intramuscular injection.
6. Having received immunoglobulin, blood, or any blood-derived product in the 3 months prior to the date of the first study vaccination or having had immunoglobulin or blood-derived product administered during the entire follow-up of the study.
7. Having received a solid organ, bone marrow, or stem cell transplant.
8. Having a history of asplenia (anatomic or functional).
9. Having any confirmed or suspected immunosuppressive or immunodeficiency condition, including a history of human immunodeficiency virus (HIV) infection.
10. Having a history of Guillain-Barré syndrome or other demyelinating disease.
11. Having a history of neurological disease, seizures, or progressive or severe neurological disorder.
12. History of malignant neoplasm or previous history of malignant neoplasm being disease-free for 5 years at the date of the first study vaccination (with the exception of basal cell carcinoma of the skin), autoimmune disease (including type 1 diabetes mellitus), liver cirrhosis and renal failure.
13. History of significant, progressive or decompensated chronic disease in the 3 months prior to the date of the first study vaccination (complicated type 2 diabetes mellitus, liver disease, kidney disease, heart disease, advanced arteriosclerotic disease or lung disease such as oxygen-dependent chronic obstructive pulmonary disease, among others).
14. Having received or using radiotherapy, chemotherapy, cytotoxic drugs, immunosuppressants or immunomodulators in the 6 months prior to the date of the first study vaccination.
15. Use of systemic corticosteroids (oral or parenteral) in the 3 months prior to the date of the first study vaccination, at an immunosuppressive dose equivalent to a dose of ≥ 20 mg of prednisone per day for ≥ 14 days or a cumulative dose of ≥ 280 mg. Topical use of corticosteroids (e.g., cream, eye drops, inhalation and intranasal sprays) is permitted, within the dosage indicated on the product label.
16. Presenting a behavioral, cognitive disorder/disorder or psychiatric illness that, in the opinion of the Investigator, may interfere with the ability to participate in the study.
17. Infection with the human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
18. Abuse of alcohol or drugs in the 12 months prior to the date of the first study vaccination, that may interfere with the ability to participate in the study.
19. Body mass index (BMI) ≥ 35 kg/m2 on the date of the first study vaccination.
20. Clinically significant abnormalities in the general physical examination.
21. Major surgery or surgery with the use of general anaesthesia planned to occur in the period from the first vaccination to the visit to assess the immune response after the last vaccination.
22. Women who are pregnant, breastfeeding or planning to become pregnant during the 30 days after the last vaccination in the study.
23. Laboratory parameter values at the screening visit equal to or greater than grade 2 will be considered as a criterion for exclusion from participation in the study.
24. Presenting any clinically significant condition or situation that, in the opinion of the Investigator, represents a risk to the participant health or may interfere with the evaluation of the study objectives, the schedule of visits, participation in or completion of the study (such as planned travel or change of residence, among others).
25. Having participated in another clinical trial involving an experimental product, with less than three months between the completion of that follow-up and the planned date of the first vaccination in this study, or plans to enter a clinical study during the period of this study.
26. Institutionalized individual (people residing in long-term care, assistance or health care institutions and deprived of liberty).

aa. Being related to or part of the research centre staff or employee directly involved in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety - Percentage of participants with solicited and unsolicited adverse events | 7 days post each vaccination.
  Percentage (%) of participants with solicited (local and systemic) and unsolicited adverse events, for each intervention group, in adults and older adults.
Safety - Percentage of solicited and unsolicited adverse events by intensity degree | 7 days post each vaccination
  Percentage of solicited and unsolicited adverse events by intensity degree for each intervention group, in adults and older adults.
Safety - Percentage of participants with solicited and unsolicited adverse reactions | 7 days post each vaccination
  Percentage of participants with solicited and unsolicited adverse reactions, for each intervention group, in adults and older adults.
Safety - Percentage of solicited and unsolicited adverse reactions by intensity degree | 7 days post each vaccination
  Percentage of solicited and unsolicited adverse reactions by intensity degree for each intervention group, in adults and older adults.
Safety - Description of solicited adverse reactions, regarding duration, time until onset and use of medication | 7 days post each vaccination
  Description of solicited adverse reactions, regarding duration, time until onset and use of medication, for each intervention group, in adults and older adults.
Immunogenicity - Seroconversion rate post second vaccination | 21 days post second vaccination
  Seroconversion rate after the second vaccination (by the hemagglutination inhibition test - HI), for each intervention group, in adults and older adults.
Immunogenicity - Seroprotection rate post second vaccination | 21 days post second vaccination
  Seroprotection rate after the second vaccination (by the hemagglutination inhibition test - HI), for each intervention group, in adults and older adults.

SECONDARY OUTCOMES:
Safety - Percentage of participants with unsolicited adverse events | 21 days post each vaccination
  Percentage of participants with unsolicited adverse events, for each intervention group, in adults and older adults.
Safety - Percentage and intensity of unsolicited adverse events | 21 days post each vaccination
  Percentage and intensity of unsolicited adverse events, for each intervention group, in adults and older adults.
Safety - Percentage of participants with unsolicited adverse reactions | 21 days post each vaccination
  Percentage of participants with unsolicited adverse reactions, for each intervention group, in adults and older adults.
Safety - Percentage and intensity of unsolicited adverse reactions | 21 days post second vaccination
  Percentage and intensity of unsolicited adverse reactions,, for each intervention group, in adults and older adults.
Percentage of participants with adverse events of special interest (AEI) | the entire follow-up of the study (6 months)
  Percentage of participants with adverse events of special interest (AEI), for each intervention group, in adults and older adults.
Safety - Percentage and intensity of the participants with adverse events of special interest (AEI) | The entire follow-up of the study (6 months)
  Percentage and intensity of the participants with adverse events of special interest (AEI), for each intervention group, in adults and older adults.
Safety - Percentage of participants with serious adverse events (SAE) | Entire follow-up of the study (6 months)
  Percentage of participants with serious adverse events (SAE), for each intervention group, in adults and older adults.
Safety - Percentage and intensity of serious adverse events (SAE) | entire follow-up of the study (6 months)
  Percentage and intensity of serious adverse events (SAE), for each intervention group, in adults and older adults.
Immunogenicity - Ratio between the Geometric Mean Titers (rGMT) of antibodies | 21 days post the first vaccination
  Ratio between the Geometric Mean Titers (rGMT) of antibodies compared to that of pre-vaccination (by the hemagglutination inhibition test - HI), for each intervention group, in adults and older adults.
Immunogenicity - Ratio between the Geometric Mean Titers (rGMT) of antibodies | 21 days post the second vaccination
  Ratio of the Geometric Mean Titers (rGMT) of antibodies, post second vaccination about that of pre-vaccination (by the hemagglutination inhibition test - HI), for each intervention group, in adults and older adults.
Immunogenicity - Seroconversion rate | 21 days post the first vaccination
  Seroconversion rate (by the hemagglutination inhibition test - HI), for each intervention group, in adults and older adults.
Immunogenicity - Geometric Mean Titers (GMT) | pre-vaccination, 21 days post the first vaccination and 21 days post the second vaccination.
  Geometric Mean Titers (GMT) pre and post-vaccination (by the hemagglutination inhibition test - HI), for each intervention group, in adults and older adults.
Immunogenicity - Seroprotection rate | pre-vaccination and 21 days post first vaccination
  Seroprotection rate pre and post-vaccination (by the hemagglutination inhibition test - HI), for each intervention group, in adults and older adults.
Immunogenicity - Ratio between the Geometric Mean Titers (rGMT) of antibodies | 21 days post the first vaccination
  Ratio between the Geometric Mean Titers (rGMT) of antibodies, pre and post-vaccination (by microneutralization test - MN), for each intervention group, in adults and older adults.
Immunogenicity - Ratio between the Geometric Mean Titers (rGMT) of antibodies | 21 days post the second vaccination
  Ratio between the Geometric Mean Titers (rGMT) of antibodies, pre and post-vaccination (by microneutralization test - MN), for each intervention group, in adults and older adults.
Immunogenicity - Seroconversion rate pre and post vaccination | 21 days post the first vaccination and 21 days post the second vaccination.
  Seroconversion rate 21 days post the first vaccination and 21 days post the second vaccination (by microneutralization test - MN), for each intervention group, in adults and older adults.
Immunogenicity - Seroprotection rate pre and post-vaccination | pre-vaccination, 21 days post the first vaccination and 21 days post the second vaccination
  Seroprotection rate pre-vaccination, 21 days after the first vaccination and 21 days after the second vaccination (by microneutralization test - MN), for each intervention group, in adults and older adults.
Immunogenicity - Geometric Mean Titers (GMT) pre and post-vaccination | pre vaccination, 21 days post the first vaccination and 21 days post the second vaccination.
  Geometric Mean Titers (GMT) pre vaccination, 21 days post the first vaccination and 21 days after the second vaccination (by the microneutralization test - MN), for each intervention group, in adults and older adults.
Immunogenicity - Estimation of rGMT between the Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) containing 7.5 mcg of HA/dose compared to that containing 15 mcg of HA/dose | 21 days post the second vaccination
  Estimation of rGMT between the Monovalent Influenza Vaccine A (H5N8) (Inactivated, Fragmented, and Adjuvanted) containing 7.5 mcg of HA/dose compared to that containing 15 mcg of HA/dose (by the hemagglutination inhibition test - HI)

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Centro de Terapias Avançadas E Inovadoras - Ct Terapias/Ufmg, Belo Horizonte, Minas Gerais
  - Plátano Centro de Pesquisa Clínica LTDA, Recife, Pernambuco
  - Fundação Faculdade Regional de Medicina de São Jose do Rio Preto - (Centro integrado de Pesquisa CIP), São José do Rio Preto, São Paulo
  - Fundação de Apoio ao Ensino, Pesquisa e Assistência do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preta da Universidade de São Paulo - (Centro de Pesquisa Clínica - S), Serrana, São Paulo
  - Centro de Pesquisas Clínicas do Hospital das Clínicas da FMUSP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akamatsu MA, Sakihara VA, Carvalho BP, de Paiva Abrantes A, Takano MAS, Adami EA, Yonehara FS, Dos Santos Carneiro P, Rico S, Schanoski A, Meros M, Simpson A, Phan T, Fox CB, Ho PL. Preparedness against pandemic influenza: Production of an oil-in-water emulsion adjuvant in Brazil. PLoS One. 2020 Jun 3;15(6):e0233632. doi: 10.1371/journal.pone.0233632. eCollection 2020. PMID 32492039
- [Background] Francis DP, Du YP, Precioso AR. Global vaccine supply. The increasing role of manufacturers from middle income countries. Vaccine. 2014 Sep 15;32(41):5259-65. doi: 10.1016/j.vaccine.2014.07.069. Epub 2014 Aug 8. PMID 25110294
- [Background] Miyaki C, Meros M, Precioso AR, Raw I. Influenza vaccine production for Brazil: a classic example of successful North-South bilateral technology transfer. Vaccine. 2011 Jul 1;29 Suppl 1:A12-5. doi: 10.1016/j.vaccine.2011.04.127. PMID 21684420
- [Background] Vanni T, Thome BC, Sparrow E, Friede M, Fox CB, Beckmann AM, Huynh C, Mondini G, Silveira DH, Viscondi JYK, Braga PE, Silva AD, Salomao MDG, Piorelli RO, Santos JP, Gattas VL, Lucchesi MBB, Oliveira MMM, Koike ME, Kallas EG, Campos LMA, Coelho EB, Siqueira MAM, Garcia CC, Miranda MD, Paiva TM, Timenetsky MDCST, Adami EA, Akamatsu MA, Ho PL, Precioso AR. Dose-sparing effect of two adjuvant formulations with a pandemic influenza A/H7N9 vaccine: A randomized, double-blind, placebo-controlled, phase 1 clinical trial. PLoS One. 2022 Oct 18;17(10):e0274943. doi: 10.1371/journal.pone.0274943. eCollection 2022. PMID 36256646